CLINICAL TRIAL: NCT04560179
Title: Phase 1 Feasibility Trial of Inhaled Tobramycin in Preterm Infants With Bronchopulmonary Dysplasia
Brief Title: Inhaled Tobramycin in BPD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Erik Allen Jensen (Other)
Collaborators: University of Florida (Other)
Responsible Party: Sponsor-Investigator, Erik Allen Jensen, Assistant Professor of Pediatrics / Attending Neonatologist, Children's Hospital of Philadelphia
Organization: Children's Hospital of Philadelphia (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 19-016800
Record Dates: First submitted 2020-09-17; First posted 2020-09-23 (Actual); Results first posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2024-12

CONDITIONS: Bronchopulmonary Dysplasia
MeSH Terms: conditions — Bronchopulmonary Dysplasia | interventions — Inhalation

STUDY DESIGN:
Intervention Model Description: 3+3 dose escalation trial.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Treatment Arm - 78mg (Experimental): The phase 1 trial will begin with a dose of 78mg. All treatment arms will administer study drug every 12 hours for up to 14 days (28 doses). Up to 6 infants in this arm will receive the 78mg dose of tobramycin solution for inhalation administered via vibrating mesh nebulizer. During the trial, infants in each treatment arm will undergo blood and tracheal aspirate sampling and respiratory mechanics measurements at pre-specified time points to assess dose safety and potential efficacy. Continuous pulse oximetry monitoring for the duration of the trial will also occur. Clinical data will also be recorded daily throughout the trial in all participants.
  Interventions: Drug: Tobramycin solution for inhalation 78mg dose
- Treatment Arm - 150mg (Experimental): If tolerability is demonstrated in the 78mg treatment arm following the 3+3 trial design, up to 6 infants will then be enrolled and receive 150mg of tobramycin solution for inhalation every 12 hours. The same monitoring procedures will be performed in this treatment arm as in the prior.
  Interventions: Drug: Tobramycin solution for inhalation 150mg dose
- Treatment Arm - 216mg (Experimental): If tolerability is demonstrated in the 150mg treatment arm following the 3+3 trial design, up to 6 infants will then be enrolled and receive 150mg of tobramycin solution for inhalation every 12 hours. The same monitoring procedures will be performed in this treatment arm as in the prior.
  Interventions: Drug: Tobramycin solution for inhalation 216mg dose
- Treatment Arm - 300mg (Experimental): If tolerability is demonstrated in the 216mg treatment arm following the 3+3 trial design, up to 6 infants will then be enrolled and receive 150mg of tobramycin solution for inhalation every 12 hours. The same monitoring procedures will be performed in this treatment arm as in the prior.
  Interventions: Drug: Tobramycin solution for inhalation 300mg dose
- Observational Arm (No Intervention): Enrolled infants who are eligible to participate in the phase-1 trial may be enrolled in an untreated observational cohort at parental discretion. This cohort will undergo collection of clinical and respiratory mechanics data for 14 days after enrollment but will not receive the study drug.

INTERVENTIONS:
Drug: Tobramycin solution for inhalation 78mg dose — Inhaled tobramycin - 78mg administered every 12 hours for 14 days.
  Arms: Treatment Arm - 78mg
Drug: Tobramycin solution for inhalation 150mg dose — Inhaled tobramycin - 150mg administered every 12 hours for 14 days.
  Arms: Treatment Arm - 150mg
Drug: Tobramycin solution for inhalation 216mg dose — Inhaled tobramycin - 216mg administered every 12 hours for 14 days.
  Arms: Treatment Arm - 216mg
Drug: Tobramycin solution for inhalation 300mg dose — Inhaled tobramycin - 300mg administered every 12 hours for 14 days.
  Arms: Treatment Arm - 300mg

SUMMARY:
This study is an open-label, phase 1, sequential dose escalation trial seeking to establish preliminary tolerability, efficacy, and pharmacokinetic data for up to 4 different doses of inhaled tobramycin administered to very preterm infants with BPD who are receiving invasive mechanical ventilation and have a pathogenic Gram-negative organism detected by tracheal aspirate culture.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female infants born <32 weeks' gestation
2. Diagnosed with BPD (use of supplemental oxygen or respiratory support at 36 weeks postmenstrual age )
3. Postmenstrual age ≥36 weeks at study enrollment
4. Treatment with invasive mechanical ventilation at enrollment without planned tracheal extubation within 7 days after enrollment
5. Tracheal aspirate culture positive for one of the following pathogenic GNR bacteria within 7 days prior to enrollment: Pseudomonas aeruginosa, Klebsiella species, Enterobacter species, Stenotrophomonas maltophilia, Escherichia coli, Acinetobacter baumannii, or Serratia marcescens
6. Parental/guardian permission (informed consent).

Exclusion Criteria:

1. Serum creatinine >0.4mg/dL within 14 days prior to enrollment
2. Congenital or acquired disease of the kidney or renal collecting system that adversely affects renal function
3. Congenital or acquired hepatobiliary disease that adversely affects liver function
4. Treatment with a systemic antibiotic within 7 days prior to enrollment
5. Treatment with a nephrotoxic medication, excluding diuretics, within 48 hours prior to enrollment
6. Treatment with a neuromuscular blocker within 48 hours prior to enrollment
7. Known intolerance to aminoglycoside antibiotics
8. Current treatment with high frequency or other oscillating mechanical ventilation
9. Presence of a cancer diagnosis
10. Maternal family history of early onset hearing loss defined as the need for an assistive hearing device prescribed before 30 years of age
11. Endotracheal tube leak >20%.
12. Any prior use of an investigational drug [as part of an FDA approved Investigational New Drug (IND) protocol].
13. A subject who, in the judgement of the Investigator, is not an appropriate candidate for this research study.

Min Age: 4 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2022-03-22 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-05-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 27 infants were enrolled into the study protocol and underwent collection of a screening tracheal aspirate culture to determine eligibility for the entry into the phase 1 drug trial. Of these 27, 16 (59%) infants had a tracheal aspirate culture positive for an eligible Gram-negative pathogen. OF these 16, all were enrolled into the phase 1 drug trial. No parents/guardians elected to enroll their child in the untreated observational arm prior to completion of all dose levels.
Period: Overall Study
Arm/Group | Treatment Arm - 78mg | Treatment Arm - 150mg | Treatment Arm - 216mg | Treatment Arm - 300mg | Observational Arm
Started | 4 | 3 | 3 | 6 | 0
Completed | 3 | 3 | 3 | 5 | 0
Not Completed | 1 | 0 | 0 | 1 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: A total of 27 infants were enrolled into the study protocol and underwent collection of a screening tracheal aspirate culture to determine eligibility for the entry into the phase 1 drug trial. Of these 27, 16 (59%) infants had a tracheal aspirate culture positive for an eligible Gram-negative pathogen. OF these 16, all were enrolled into the phase 1 drug trial. No parents/guardians elected to enroll their child in the untreated observational arm prior to completion of all dose levels.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Arm - 78mg | Treatment Arm - 150mg | Treatment Arm - 216mg | Treatment Arm - 300mg | Observational Arm | Total
Number analyzed (Participants) | 4 | 3 | 3 | 6 | 0 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 3 | 3 | 6 | 0 | 16
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 2 | 2 | 0 | 7
  Male | 3 | 1 | 1 | 4 | 0 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 0 | 1 | 0 | 4
  Not Hispanic or Latino | 1 | 3 | 3 | 5 | 0 | 12
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 3 | 3 | 2 | 0 | 11
  White | 1 | 0 | 0 | 1 | 0 | 2
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 3 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 3 | 6 |  | 16

OUTCOME MEASURES:

1. Primary Outcome: Elevated Serum Tobramycin Trough or Creatinine or Severe Adverse Event
Description: Trough serum tobramycin level (measured 11 hours after the administered dose) ≥1mcg/mL; increase in serum creatinine level by ≥0.3mg/dL above pre-trial baseline; increase in serum creatinine level >1.5-fold above pre-trial baseline; urine output <0.5mL/kg/hr for 12 consecutive hours; or any serious adverse event possibly attributable to the study drug
Time Frame: Any time during the 14-day trial
Population: No infants were enrolled into the observational arm. 1 of the 16 enrolled infants (treatment arm - 78mg) was withdrawn early from the trial by the medical team and was not assessed for this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm - 78mg | Treatment Arm - 150mg | Treatment Arm - 216mg | Treatment Arm - 300mg | Observational Arm
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 0
Participants | 0 | 0 | 0 | 1 | 0

2. Secondary Outcome: New Onset or Worsened Coughing Associated With a Change in Respiratory Status (SpO2 <80% for >10 Seconds; Need for Increase in FiO2 by >20%)
Time Frame: Any time during the 14-day trial
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm - 78mg | Treatment Arm - 150mg | Treatment Arm - 216mg | Treatment Arm - 300mg | Observational Arm
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 0
Participants | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Obstruction of the Endotracheal Tube Requiring Tube Replacement
Time Frame: Any time during the 14-day trial
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm - 78mg | Treatment Arm - 150mg | Treatment Arm - 216mg | Treatment Arm - 300mg | Observational Arm
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 0
Participants | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Unplanned Tracheal Extubation
Time Frame: Any time during the 14-day trial
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm - 78mg | Treatment Arm - 150mg | Treatment Arm - 216mg | Treatment Arm - 300mg | Observational Arm
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 0
Participants | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Desaturation (SpO2 <80% for >10 Seconds) During Administration of Inhaled Tobramycin
Time Frame: Any time during the 14 day trial
Population: No infants were enrolled into the observational arm. Infants who were screened but not eligible did not receive study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Screened But Not Eligible: Enrolled infants who did not have evidence of a Gram-negative bacteria present on a prospective tracheal aspirate culture obtained for this trial and thus were not eligible to receive study drug.
Arm/Group | Treatment Arm - 78mg | Treatment Arm - 150mg | Treatment Arm - 216mg | Treatment Arm - 300mg | Observational Arm | Screened But Not Eligible
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 0 | 0
Participants | 3 | 0 | 1 | 0 | 0 | 0

6. Secondary Outcome: Pre-discharge Failed Audiology Examination
Time Frame: up to 1 year of age
Population: 14 of the 16 phase 1 trial participants were assessed for failed audiology examination. The remaining two died prior to testing.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm - 78mg | Treatment Arm - 150mg | Treatment Arm - 216mg | Treatment Arm - 300mg | Observational Arm
Number analyzed (Participants) | 3 | 3 | 3 | 5 | 0
Participants | 1 | 1 | 0 | 1 | 0

7. Secondary Outcome: New Intra-patient Microbial Resistance to Tobramycin During the Primary Hospitalization
Time Frame: up to 1 year of age
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm - 78mg | Treatment Arm - 150mg | Treatment Arm - 216mg | Treatment Arm - 300mg | Observational Arm
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 0
Participants | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Change in Tracheal Aspirate Pathogenic Bacterial Colony Forming Unit (CFU) Counts Measured by Quantitative Culture
Time Frame: During the 14-day trial
Population: CFU counts were not measured by the microbiology lab on tracheal aspirate samples; only presence/absence of pathogens was recorded owing to variable consistency of sputum samples. No infants were enrolled into the observational arm.
Arm/Group | Treatment Arm - 78mg | Treatment Arm - 150mg | Treatment Arm - 216mg | Treatment Arm - 300mg | Observational Arm
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Change in the Fraction of Inspired Oxygen (FiO2), Ventilator Mean Airway Pressure (MAP), and Respiratory Severity Score (MAP x FiO2)
Time Frame: During the 14-day trial
Reporting Status: Not Posted, anticipated posting 2025-12

10. Secondary Outcome: Change in Intermittent Hypoxemia (SpO2<80% Lasting >/=10s), Prolonged Hypoxemia (SpO2<80% Lasting >1min), and Daily Proportion of Time in Hypoxemia
Time Frame: During the 14-day trial
Reporting Status: Not Posted, anticipated posting 2025-12

11. Secondary Outcome: Change in Tracheal Aspirate Cytokine Levels, Neutrophil to Total WBC Ratio, and Patterns in the Airway Microbiome
Time Frame: During the 14-day trial
Reporting Status: Not Posted, anticipated posting 2025-12

12. Secondary Outcome: Change in Dynamic Lung Compliance, Airway Resistance, Peak Expiratory Flow, and Carbon Dioxide (CO2) Elimination
Time Frame: During the 14-day trial
Reporting Status: Not Posted, anticipated posting 2025-12

ADVERSE EVENTS:
Time Frame: During the 14 day drug trial and continuing until hospital discharge
Description: Adverse event data was not captured on infants who were screened but not enrolled into the drug trial.
Arm/Group | Treatment Arm - 78mg | Treatment Arm - 150mg | Treatment Arm - 216mg | Treatment Arm - 300mg | Observational Arm | Screened But Not Eligible
All-Cause Mortality (participants affected / at risk) | 2/4 | 0/3 | 1/3 | 1/6 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3 | 0/3 | 0/6 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/4 | 1/3 | 1/3 | 1/6 | 0/0 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm - 78mg (N=4) | Treatment Arm - 150mg (N=3) | Treatment Arm - 216mg (N=3) | Treatment Arm - 300mg (N=6) | Observational Arm (N=0) | Screened But Not Eligible (N=0)
Desturation episode outside of study drug administration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) — Episodes of desaturation (SpO2<80%) lasting longer than 30 seconds that is possibly/probably related to study drug administration

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-20): https://cdn.clinicaltrials.gov/large-docs/79/NCT04560179/Prot_SAP_000.pdf